CLINICAL TRIAL: NCT03337399
Title: Randomized Trial of Stepped Palliative Care Versus Early Integrated Palliative Care in Patients With Advanced Lung Cancer
Brief Title: Stepped Palliative Care Versus Early Integrated Palliative Care in Patients With Advanced Lung Cancer
Acronym: STEP PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Temel, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-471; R01CA215188 (NIH)
Record Dates: First submitted 2017-11-06; First posted 2017-11-09 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepped PC (Experimental): * Patients will receive Stepped PC
  * During step 1, patients will be scheduled to meet with the outpatient PC clinician within four weeks of study enrollment and after they are admitted to the hospital or have a change in their cancer treatment
  * Patients will complete the Functional Assessment of Cancer Therapy-Lung (FACT-L) to monitor their quality of life every six weeks and if their quality of life deteriorates substantially, they will "step up" to step 2 of the protocol
  * Patients who transition to step 2 will then meet with the PC clinician at least every four weeks for the remainder of their illness
  Interventions: Other: Stepped PC
- Early Integrated PC (Experimental): * Patients will receive Early Integrated PC
  * Patients will meet with the PC clinician within four weeks of enrollment and at least every four weeks throughout their course of illness
  Interventions: Other: Early Integrated PC

INTERVENTIONS:
Other: Stepped PC — Palliative Care is involvement of a team of clinicians that specialize in lessening (or "palliating") many of these distressing physical and emotional symptoms and in helping patients and their family cope with a serious illness improves patients' and their loved ones' experience with their cancer
  Arms: Stepped PC
Other: Early Integrated PC — Palliative Care is involvement of a team of clinicians that specialize in lessening (or "palliating") many of these distressing physical and emotional symptoms and in helping patients and their family cope with a serious illness improves patients' and their loved ones' experience with their cancer
  Arms: Early Integrated PC

SUMMARY:
This research study is evaluating ways to provide palliative care to patients who have recently been diagnosed with lung cancer

DETAILED DESCRIPTION:
Patients with serious cancers, like advanced lung cancer, often experience physical symptoms, such as pain or shortness of breath. In addition, both patients and their loved ones (family and friends) often feel worried or sad about their cancer diagnosis.

Research has shown that early involvement of a team of clinicians that specialize in lessening (or "palliating") many of these distressing physical and emotional symptoms and in helping patients and their family cope with a serious illness improves patients' and their loved ones' experience with their cancer. This team is called "palliative care," and consists of physicians and advanced practice nurses (or "nurse practitioners") who work closely and collaboratively with your oncology team to care for the participant and the participant's loved ones. Research shows that when the palliative care team works closely with the oncology team to care for patients with advanced cancer, they may have better symptom control, quality of life, and mood and their loved ones feel less distressed.

This study will compare two different strategies for scheduling participant's visits with the palliative care clinician. The first strategy is to schedule the participant to meet with the palliative care clinician regularly each month. The investigators call this strategy "early integrated palliative care".

The second strategy is to schedule the participant to meet with the palliative care clinician after the participant is admitted to the hospital or if the participant's oncology team needs to change the participant cancer treatment, as these are times when the participant is likely to have health issues that the palliative care clinician can help with. The investigators will also monitor the participant's quality of life regularly. If the study team determines that the participant quality of life worsens, the investigators will increase the frequency of the participant's visits with the palliative care clinician to monthly appointments. The investigators call this strategy "stepped palliative care" because the investigators step up the frequency of the participant palliative care visits if the participant's quality of life worsens during the participant cancer treatment.

No matter which strategy the participant is taking part in, the participant will still be able to request additional palliative care visits outside of the study schedule if the participant feel they need them.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with advanced non-small cell lung cancer, small cell lung cancer, or mesothelioma, being treated with non-curative intent, and informed of advanced disease within the prior twelve weeks
* Eastern Cooperative Oncology Group (ECOG) Performance Status from 0 (asymptomatic) to 2 (symptomatic and in bed <50% of the day)
* The ability to read and respond to questions in English or Spanish
* Primary cancer care at one of the three participating sites
* Age > 18 years

Exclusion Criteria:

* Already receiving outpatient PC or hospice services
* Cognitive or psychiatric conditions as determined by the treating oncologist to prohibit study consent or participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Temel, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Temel JS, Jackson VA, El-Jawahri A, Rinaldi SP, Petrillo LA, Kumar P, McGrath KA, LeBlanc TW, Kamal AH, Jones CA, Rabideau DJ, Horick N, Pintro K, Gallagher Medeiros ER, Post KE, Greer JA. Stepped Palliative Care for Patients With Advanced Lung Cancer: A Randomized Clinical Trial. JAMA. 2024 Aug 13;332(6):471-481. doi: 10.1001/jama.2024.10398. PMID 38824442
- [Derived] Petrillo LA, El-Jawahri A, Heuer LB, Post K, Gallagher ER, Trotter C, Elyze M, Vyas C, Plotke R, Turk YR, Han J, Temel JS, Greer JA. Health-Related Quality of Life and Depression Symptoms in a Cross Section of Patients with Advanced Lung Cancer before and during the COVID-19 Pandemic. J Palliat Med. 2022 Nov;25(11):1639-1645. doi: 10.1089/jpm.2022.0049. Epub 2022 May 19. PMID 35588200
- [Derived] Post KE, Heuer LB, Kamal AH, Kumar P, Elyze M, Griffith S, Han J, Friedman F, Jackson A, Trotter C, Plotke R, Vyas C, Jackson V, Rabideau DJ, Greer JA, Temel JS. Study protocol for a randomised trial evaluating the non-inferiority of stepped palliative care versus early integrated palliative care for patients with advanced lung cancer. BMJ Open. 2022 Feb 10;12(2):e057591. doi: 10.1136/bmjopen-2021-057591. PMID 35144954

RESULTS

PARTICIPANT FLOW:
Groups:
- Stepped PC: * Patients will receive Stepped PC
  * During step 1, patients will be scheduled to meet with the outpatient PC clinician within four weeks of study enrollment and after they are admitted to the hospital or have a change in their cancer treatment
  * Patients will complete the Functional Assessment of Cancer Therapy-Lung (FACT-L) to monitor their quality of life every six weeks and if their quality of life deteriorates substantially, they will "step up" to step 2 of the protocol
  * Patients who transition to step 2 will then meet with the PC clinician at least every four weeks for the remainder of their illness
  Stepped PC: Palliative Care is involvement of a team of clinicians that specialize in lessening (or "palliating") many of these distressing physical and emotional symptoms and in helping patients and their family cope with a serious illness improves patients' and their loved ones' experience with their cancer
- Early Integrated PC: * Patients will receive Early Integrated PC
  * Patients will meet with the PC clinician within four weeks of enrollment and at least every four weeks throughout their course of illness
  Early Integrated PC: Palliative Care is involvement of a team of clinicians that specialize in lessening (or "palliating") many of these distressing physical and emotional symptoms and in helping patients and their family cope with a serious illness improves patients' and their loved ones' experience with their cancer
Period: Overall Study
Arm/Group | Stepped PC | Early Integrated PC
Started | 250 | 257
Completed | 250 | 257
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stepped PC | Early Integrated PC | Total
Number analyzed (Participants) | 250 | 257 | 507
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (9.2) | 66.1 (11.1) | 66.5 (10.2)
Sex/Gender, Customized [Number; unit: participants]
  Woman | 130 | 130 | 260
  Man | 120 | 126 | 246
  Other | 0 | 0 | 0
  Missing | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 28 | 57
  White | 215 | 212 | 427
  More than one race | 0 | 5 | 5
  Unknown or Not Reported | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 250 | 257 | 507
Functional Assessment of Cancer Therapy - Lung [Mean (Standard Deviation); unit: units on a scale] — Range 0-136 with higher scores indicating better quality of life
  units on a scale | 93.6 (19.4) | 95.7 (19.7) | 94.63 (19.60)

OUTCOME MEASURES:

1. Primary Outcome: Patient-reported Quality of Life
Description: Quality of life as measured by the Functional Assessment of Cancer Therapy-Lung Range 0-136 with higher scores indicating better quality of life
Time Frame: 24 Weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stepped PC | Early Integrated PC
Number analyzed (Participants) | 250 | 257
score on a scale | 100.62 [98.10 to 103.14] | 97.75 [95.18 to 100.33]
Statistical Analysis 1: Comparison: Stepped PC vs Early Integrated PC; The difference in week 24 means between groups was estimated using a linear regression model adjusted for baseline FACT-L score; Test type: Non-Inferiority — Non-inferiority of stepped PC was established if the lower one-sided 95% confidence limit for the estimated difference in means was greater than the pre-specified margin of -4.5 points, which corresponds to the one-sided 5% significance level test against this margin; p < 0.05, Regression, Linear; Mean Difference (Final Values) = 2.9, 95% CI 1-sided [lower limit -.01]

2. Secondary Outcome: Proportion of Patients Who Self-report Discussing Their End of Life Care Preferences With Their Clinicians
Description: Compare the proportion of patients who report that they discussed their end-of-life care preferences with their clinicians based on a single item from the perceptions of prognosis and treatment questionnaire (PTPQ). The PTPQ includes an item that measures patient report of communication about their wishes if they were dying (yes vs. no).
Time Frame: 48 weeks (or last assessment prior to death if before 48 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Stepped PC | Early Integrated PC
Number analyzed (Participants) | 190 | 187
Participants | 58 | 62
Statistical Analysis 1: Comparison: Stepped PC vs Early Integrated PC; Non-inferiority of stepped PC in the proportion reporting patient-clinician communication about end-of-life care at each patient's final follow-up assessment was evaluated using a binomial generalized linear model with identity link and a one-sided test against the pre-specified margin of -10%; Test type: Non-Inferiority — Pre-specified margin of -10%; p < 0.15, Regression, Linear — We used a false discovery rate (FDR) control approach to interpret the results of significance tests of the three secondary outcomes with an FDR of 0.15; Estimated Proportions = -2.6, 95% CI 1-sided [lower limit -10.4]

3. Secondary Outcome: Length of Stay in Hospice
Description: Length of stay in hospice as collected per medical record review
Time Frame: From hospice enrollment until death during study period (i.e. 12-month follow up)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Stepped PC | Early Integrated PC
Number analyzed (Participants) | 159 | 161
days | 19.5 (4.3) | 34.6 (4.2)
Statistical Analysis 1: Comparison: Stepped PC vs Early Integrated PC; Among patients who died, non-inferiority of stepped PC in the mean length of stay in hospice was assessed using linear regression and a one-sided test against the pre-specified margin of -7 days, based upon published quality metrics; Test type: Non-Inferiority — Pre-specified margin of -7 days; p = 0.15, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Median Difference (Final Values) = -15.2, 95% CI 1-sided [lower limit -25.1]

4. Secondary Outcome: Palliative Care Resource Utilization
Description: Mean number of palliative care visits
Time Frame: week 24
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Stepped PC | Early Integrated PC
Number analyzed (Participants) | 250 | 257
days | 2.4 (0.2) | 4.7 (0.1)
Statistical Analysis 1: Comparison: Stepped PC vs Early Integrated PC; The difference between groups in the mean number of outpatient PC visits per patient by week 24 was assessed using linear regression and a two-sided superiority test; Test type: Superiority; p = 0.15, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Median Difference (Final Values) = -2.3, 95% CI 2-sided [-2.7 to -1.8]

5. Other Pre Specified Outcome: Cost-effectiveness
Description: Cost effectiveness as assessed by data collection from the medical record, hospital cost accounting systems, and patient report as per the EuroQOL
Time Frame: up to 5 years
Reporting Status: Not Posted, anticipated posting 2025-12

6. Other Pre Specified Outcome: Patients' Prognostic Understanding
Description: Perception of Treatment and Prognosis Questionnaire (PTPQ)
Time Frame: last assessment collected during study or prior to death
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Health Care Utilization
Description: Healthcare utilization as measured the means and proportion of patients who experience emergency department visits, hospital admission, and chemotherapy administration at the end of life between the two groups.
Time Frame: prior to death or end of study period
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: Up to 12 months post enrollment
Description: No serious or other (non-serious) adverse events were collected or monitored in this supportive care trial. As a result, the total number of participants at risk for adverse events is zero since this was not monitored in this supportive care trial.
Arm/Group | Stepped PC | Early Integrated PC
All-Cause Mortality (participants affected / at risk) | 161/250 | 164/257
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT03337399/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT03337399/SAP_001.pdf